CLINICAL TRIAL: NCT05944068
Title: The Effects of a Mindfulness Based Intervention on IBD Disability
Acronym: EMBODY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S67980
Record Dates: First submitted 2023-06-23; First posted 2023-07-13 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: EMBODY (Effects of a Mindfulness Based interventiOn on ibD disabilitY) will be a prospective, randomized-controlled, monocentric, superiority trial using a waiting list with treatment as usual as control arm. Half of the patients will immediately start the mindfulness based intervention (early intervention group). In the other half, there will be a waiting time of 6 months before starting the mindfulness based intervention (late intervention or control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention group (Experimental): This group will receive the intervention immediately after baseline.
  Interventions: Behavioral: midfulness training
- Late intervention group (Other): This group will receive the intervention 6 months after baseline, in psychological studies called the waiting list group
  Interventions: Behavioral: midfulness training

INTERVENTIONS:
Behavioral: midfulness training — For this study we chose for a mindfulness based intervention. Mindfulness is defined as the ability to notice and observe details about one's present internal and external environment with the goal of non-judgemental and non-elaborative awareness of cognitions, emotions and physical sensations. The goal of the mindfulness intervention will be to teach patients a way of coping with negative emotions without acting on them, letting patients take control of their disease related behaviour and come to better disease acceptance. Where medical treatments fail to take away all disabling symptoms, psychological interventions like mindfulness could offer patients a coping method through which symptoms are experienced as less disabling and patients regain their quality of life. This research may further strengthen the need for a multidisciplinary approach in patients with Crohn's disease.

SUMMARY:
EMBODY (Effects of a Mindfulness Based interventiOn on ibD disabilitY) aims to evaluate the effects of a mindfulness based intervention on a broad number of disease related disability dimensions in patients with Crohn's disease (abdominal pain, regulation defecation, joint pain, energy, emotions, body image, interpersonal interactions, education and work, sexual function, sleep). Besides, the investigators will measure the effect of the intervention on depression, anxiety, stress, disease acceptance and perceived control as well as (biomarkers of) disease activity. It will be a prospective, randomized-controlled, monocentric, superiority trial using a waiting list with treatment as usual as control arm. Half of the patients will immediately start the mindfulness based intervention (early intervention group). In the other half, there will be a waiting time of 6 months before starting the mindfulness based intervention (late intervention or control group). Clinical disease activity (two-item patient reported outcome (PRO2)), faecal calprotectin and C-reactive protein (CRP) will be collected throughout the trial (pre-, during and post-intervention). The investigators will measure IBD-related disability through the IBD-Disk, a tool for assessing the impact of the disease on ten different dimensions of everyday life dimensions. Depression, anxiety and Stress will be investigated via the Depression Anxiety Stress Scale Short Form (DASS21). Disease acceptance and perceived control will be measured using the Subjective Health Experience (SHE) model. Evolution of the different variables will be compared between both groups (ANOVA).

DETAILED DESCRIPTION:
Crohn's disease (CD), next to ulcerative colitis (UC), is an inflammatory bowel disease (IBD) and causes chronic inflammation of the intestine. Patients suffer from chronic or relapsing symptoms as diarrhea, rectal blood loss, abdominal pain, nausea and weight loss. Next to physical symptoms, a large number of Crohn's disease patients present psychological distress, due to the large impact the disease has on daily life functioning. Depression and anxiety, as well as chronic fatigue are more prevalent in patients with Crohn's disease compared to healthy controls. The disease also significantly affects other biopsychosocial factors, including interpersonal relationships, educational or work-related activities, body image, sleep and sexual functioning. The impact of the disease on these factors translates to the amount of disease related disability Crohn's patients experience during daily life.

With this study, the investigators will evaluate the effects of a mindfulness based psychological intervention on a broad number of disease related disability factors in patients with Crohn's disease. Besides, they would like to measure the effect of the intervention on perceived stress, disease acceptance and perceived control as well as (biomarkers of) disease activity.

In many patients with Crohn's disease, objective markers of inflammation deviate from subjective health outcomes. For instance, patients may report impairing symptoms even in the absence of active disease, often resulting in comorbid psychological distress. Nearly 80% of those with active disease and 50% of those with inactive IBD report substantial fatigue that impairs their health related quality of life (HRQoL). Next to fatigue, other life domains measured by the IBD Disk, a short instrument that can clinically be used as a measure of patient-reported IBD-related disability, are abdominal pain, regulated defecation, interpersonal interactions, education and work, sleep, emotions, body image, sexual functions, and joint pain.

The relation between IBD and stress is bidirectional. Not only are patients with IBD who are experiencing symptoms more likely to have higher levels of perceived stress, but perceived stress also has a strong and consistent association with concurrent and subsequent IBD symptoms. Furthermore, the intervention of choice (mindfulness) was originally developed as a stress reduction method. Depression and anxiety are also more prevalent in the IBD population compared to healthy controls. But not only does the disease influence mental health, mental health will also affect disease activity. A study by Gracie et al. documented a nearly sixfold increase in risk for anxiety symptoms in those with normal anxiety levels but active IBD at baseline. The same study showed a twofold increase in risk of IBD flares, need for steroids and escalation therapy in those with higher anxiety but quiescent IBD activity at baseline. Hence, the investigators chose to also measure depression, anxiety and stress by means of the Depression Anxiety Stress Scale Short Form (DASS21).

Two other important psychological determinants of subjective health are disease acceptance and perceived control over the disease, both integrated in the SHE model. The definition given by Bloem and Stalpers for disease acceptance is "the feeling by the individual that his health condition and the possible constraints on functioning resulting from it, are acceptable and fitting for him as a person" and for perceived control "the belief of the individual that his health condition, in the individual's perception, can be influenced or controlled by himself or by others".

For this study the investigators chose for a mindfulness based intervention. Mindfulness is defined as the ability to notice and observe details about one's present internal and external environment with the goal of non-judgemental and non-elaborative awareness of cognitions, emotions and physical sensations. This allows for reflective (taking time for reflecting) versus reflexive (resulting from behavioral reflexes) reactions to situations or feelings. Mindfulness is achieved through a standard practice, including meditation, body scan practices, yoga and guided focus on different body parts.

Baer et al. proposed five mechanisms by which mindfulness might work to improve symptoms and mood: (1) exposure, by encouraging patients to experience and accept unpleasant sensations without avoidance, (2) cognitive change, by shifting the conceptualization of negative thinking from "reflections of truth" to "just thoughts", (3) self-management, by improving coping skills through enhancing awareness of thoughts, emotions and sensations, (4) relaxation, by indirectly reducing physical tension and autonomic arousal, and (5) acceptance, by promoting non-judgemental awareness of one's own personal experience and reducing maladaptive behaviours aimed at changing the experience.

The goal of the mindfulness intervention will be to teach patients a way of coping with negative emotions without acting on them, letting patients take control of their disease related behaviour and come to better disease acceptance. Where medical treatments fail to take away all disabling symptoms, psychological interventions like mindfulness could offer patients a coping method through which symptoms are experienced as less disabling and patients regain their quality of life. This research may further strengthen the need for a multidisciplinary approach in patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant has been obtained prior to any screening procedures
2. Males and females 18-80 years old.
3. Patients with a diagnosis of Crohn's disease based on radiology, endoscopy and/or histology
4. Patients with more than one year of follow-up since diagnosis
5. Patients having internet or smartphone access
6. Patients being fluent in Dutch

Exclusion Criteria:

1. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
2. Patients that initiated a new IBD medication (steroids, thiopurines, methotrexate, biologicals or small molecules) in the past three months
3. Patients in whom a major surgery or acute surgery with hospitalization can be expected during the complete study period
4. Patients with a present or past psychiatric disease diagnosis (psychosis, bipolar disease, substance abuse)
5. Patients using psychotropic medication
6. Patients with former experience of mindfulness training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The median change in the IBD-related disability index by month 3 | 6 months
  This study will evaluate if a mindfulness based intervention can improve IBD-related disability, measured through the IBD Disk. Patients are asked to rate each item on a scale from 0 to 10 (0 = absolutely disagree, 10 = absolutely agree), resulting in a total score ranging from 0 to 100. A higher score represents higher IBD-related disability.

SECONDARY OUTCOMES:
The median change in separate components of the IBD-related disability index, perceived stress, perceived control and disease acceptante by month 3 | 6 months
  The median change in the seperate components of the IBD-related disability index by month 3.
  Each item is rated on a scale from 0 to 10 (0 = absolutely disagree, 10 = absolutely agree). A higher score represents higher IBD-related disability.
  The median change in the depression/anxiety/stress scale of the DASS21 by month 3. Each of the three scales contains 7 items. Items are rated on 4-point severity/frequency scales. Higher scores represent higher probability of depression, anxiety and/or stress.
  The median change in the disease acceptance/perceived control component of the SHE model by month 3. The SHE model contains 6 questions with a scale from 1 to 7 (1=fully agree, 7=fully disagree). Higher scores represent higher perceived control/acceptance.

OTHER OUTCOMES:
Evolution of C-reactive protein and fecal calprotectin over time | 12 months
  Evolution of CRP over time. Evolution of faecal calprotectin over time.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No